CLINICAL TRIAL: NCT01990001
Title: Randomized Trial of Provider-Assisted Versus Patient-Initiated Enrollment in the Bedsider.Org Online Contraceptive Reminder Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: American College of Obstetricians and Gynecologists (Other)
Responsible Party: Principal Investigator, Ashlyn H. Savage, MD, Assistant Professor of Obstetrics and Gynecology, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Besider
Record Dates: First submitted 2013-11-11; First posted 2013-11-21 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2013-11

CONDITIONS: Contraceptive Adherence and Continuation
Keywords: contraception, adherence, medication reminder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Office enrollment in the online contraceptive reminder system (Experimental): Members of this arm were enrolled in the reminder system during their visit.
  Interventions: Other: enrollment in online reminder system
- Control (No Intervention): Members in the control group were not enrolled in the reminder system

INTERVENTIONS:
Other: enrollment in online reminder system — Study personnel enrolled members in the online reminder system during their office visit.
  Arms: Office enrollment in the online contraceptive reminder system

SUMMARY:
The broad objective of this research is to determine whether a quick, simple intervention will increase utilization of contraceptive reminders and adherence to short-term contraceptive regimens. Such an intervention could be implemented easily with no additional resources into a busy clinical practice.

DETAILED DESCRIPTION:
The specific aims of the study are to:

1. Measure the difference in reminder utilization over three months between patients who are assisted with initiating the reminder system during their office visit versus those who are encouraged to self-initiate after the visit.
2. Assess whether provider-assisted enrollment in the online reminder system improves adherence to a short-term contraceptive regimen compared to self- initiated enrollment after the visit.

ELIGIBILITY:
Inclusion Criteria:

1. Female, 18-29 years old
2. Prescribed one of the following birth control:

   Oral contraceptive pills, vaginal ring, transdermal patch, or Depo Provera
3. Able to provide consent
4. Have regular access to a computer, Ipad, or a hand-held device such as a smartphone.
5. Women must be able to read and speak English(Bedsider website in not translated into Spanish)

Exclusion Criteria:

1. Male
2. Over the age of 30 years old
3. Non-English Speaking
4. Limited or no access to computer, Ipad or hand-held device(smartphone)

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients using the online reminder tool three months after enrollment | 3 months
  Measure the difference in reminder utilization over three months between patients who are assisted with initiating the reminder system during their office visit versus those who are encouraged to self-initiate after the visit. The primary outcome, which is proportion of reminder users, will be assessed three months after enrollment

SECONDARY OUTCOMES:
Assess whether provider-assisted enrollment in the online reminder system improves adherence to a short-term contraceptive regimen compared to self- initiated enrollment after the visit. | 3 months
  Assess whether provider-assisted enrollment in the online reminder system improves adherence to a short-term contraceptive regimen compared to self- initiated enrollment after the visit. This data will be collected three months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Ashlyn Savage, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- MUSC Women's Health- Cannon, Charleston, South Carolina, United States